CLINICAL TRIAL: NCT06029660
Title: AAA-SHAPE Pivotal Trial: Abdominal Aortic Aneurysm Sac Healing and Prevention of Expansion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shape Memory Medical, Inc. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD 1029
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized, open-label trial.
Masking Description: Subjects will be blinded to the treatment arm prior to the index procedure; after the procedure, they will be unblinded prior to discharge to prevent unintentional unblinding due to imaging
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Treatment Arm: Subjects in the treatment arm will have both an EVAR device and IMPEDE-FX RapidFill implants inserted.
  Interventions: Device: IMPEDE-FX RapidFill Implants; Procedure: EndoVascular Aneurysm Repair
- Control (Active Comparator): Control Arm: Subjects in the control arm will only have an EVAR device implanted.
  Interventions: Procedure: EndoVascular Aneurysm Repair

INTERVENTIONS:
Device: IMPEDE-FX RapidFill Implants — Filling of the available flow lumen within the AAA sac with IMPEDE-FX RapidFill Implants
  Arms: Treatment
Procedure: EndoVascular Aneurysm Repair — Standard EVAR repair of abdominal aortic aneurysms using a commercially available stent.
  Other Names: EVAR

SUMMARY:
To determine the safety and effectiveness of IMPEDE-FX RapidFill to increase the percentage of subjects with shrinkage of the abdominal aortic aneurysm sac when used as an adjunct to on-label endovascular aneurysm repair (EVAR) stent graft treatment in trial subjects considered candidates for elective EVAR.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. A candidate for elective EVAR of an infrarenal fusiform aortic aneurysm ≥5.5 cm in diameter in men and ≥5.0 cm in women;
3. Thrombus burden (percentage of the AAA sac occupied by thrombus) <50%, based on pre-procedure CTA
4. Maximum Lumen diameter within the AAA sac of ≥40mm.
5. The predicted minimum number of IMPEDE-FX RapidFill Implants for the subject is ≤200.

Exclusion Criteria:

General

1. An inability to provide informed consent.
2. Enrolled in another clinical study that could interfere with the outcomes being studied in this trial.
3. Unable or unwilling to comply with study follow-up requirements.
4. Prisoner or member of other vulnerable population

Anatomical

1. Concomitant iliac artery ectasia or aneurysm
2. Vascular disease and/or anatomy that preclude the safe access and positioning of a catheter to deliver the investigational product into the AAA sac.
3. Ruptured, leaking, inflammatory or mycotic (infected) aneurysm.
4. Connective tissue disorder (e.g., Marfan's syndrome)
5. Aneurysmal disease of the descending thoracic aorta
6. Excessive calcification at the aortic bifurcation to common/internal iliac bifurcation, that might lead to access difficulties

EVAR/Procedural

1. Use of aortic stent grafts other than the Gore Excluder AAA Endoprosthesis, Gore Excluder Conformable AAA Endoprosthesis, Cook Zenith Flex AAA Endovascular Graft, Medtronic Endurant II and Endurant IIs Stent Graft, or the Terumo TREO Stent Graft to treat the AAA
2. Use of an aortic stent graft other than those specified1 for a particular site
3. Planned use of the chosen stent graft outside its instructions for use (IFU)
4. Use of fenestrated stent grafts or chimney techniques
5. Use of the Heli-FX EndoAnchor system
6. Use of embolic devices other than the investigational product to embolize the AAA sac
7. Use of embolic products to prophylactically or concomitantly embolize the inferior mesenteric artery, lumbar arteries, renal accessory arteries, or internal iliac arteries
8. Inability to land the distal-most portion of the EVAR stent graft limbs, including extensions, above the internal iliac arteries

Medical History/Conditions

1. Coagulopathy or uncontrolled bleeding disorder
2. Serum creatinine level >2.5 mg/dL
3. Cerebrovascular accident within 3 months prior to the procedure
4. Myocardial infarction and/or major heart surgery within 3 months prior to the procedure
5. Atrial fibrillation that is not well rate controlled
6. Life expectancy of <2 years post-procedure
7. Known hypersensitivity or contraindication to platinum, iridium, or polyurethane.
8. Have active infection at the time of the index procedure documented by pain, fever, drainage, positive culture, or leukocytosis (WBC >11,000/mm3)
9. A condition that inhibits radiographic visualization during the implantation procedure
10. History of allergy to contrast medium that cannot be managed medically, or subject is unable to have a CT with contrast for any reason.
11. Uncontrolled co-morbid medical condition, including mental health issues, that would adversely affect participation in the trial
12. Pregnant or lactating female: for females of child-bearing potential, based on a positive pregnancy test within 7 days prior to the procedure or refusal to use a medically accepted method of birth control for the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint : AAA Sac Regression at 1 year | 1 year
  The percentage of subjects showing regression, defined as sac volume reduction of ≥10% at 1 year (in comparison to the 30 day CT), and no AAA-related intervention through 1 year.
Primary Safety Endpoint : Major Adverse Event (MAE) Rate through 30 days | 30 days
  Freedom from the following through 30 days post-index procedure:
  * Major adverse events (MAEs) which include the following: all-cause mortality, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, stroke, procedural blood loss >1000 mL.
  * AAA-rupture or AAA-perforation
  * Conversion to Open Repair

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schermerhorn, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (45):
- United States (37):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Honor Health, Scottsdale, Arizona
  - USC Keck, Los Angeles, California
  - San Diego VA Medical Center, San Diego, California
  - Delray Medical Center, Delray Beach, Florida
  - Orlando Health, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Maine Medical, Portland, Maine
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - VA Ann Arbor Healthcare, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University at Buffalo, Buffalo, New York
  - Buffalo VA Western New York, Buffalo, New York
  - NYU Langone, New York, New York
  - Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook Medicine, Stony Brook, New York
  - TriHealth Heart Institute, Cincinnati, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - Vanderbilt University, Nashville, Tennessee
  - Houston Methodist, Houston, Texas
  - Baylor Scott and White, Plano, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Schar Heart and Vascular, Falls Church, Virginia
  - Sentara Norfolk General, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Marie Lannelongue Hospital, Paris, Le Plessis-Robinson, France
- Netherlands (4):
  - Rijnstate Hospital, Arnhem, Gelderland
  - ETZ Elisabeth, Tilburg, Tilburg
  - Amsterdam UMC, Amsterdam
  - Erasmus Medical Center, Rotterdam
- New Zealand (2):
  - Auckland City Hospital, Auckland, Auckland
  - Waikato Hospital, Hamilton
- St Georges University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No